CLINICAL TRIAL: NCT05925426
Title: Defining The Quality Of Intraoperatively Salvaged Blood For Deformity Surgery
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 22-00406
Record Dates: First submitted 2023-06-22; First posted 2023-06-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Spinal Deformity
Keywords: Red Blood Cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The actual quality of Red Blood Cells (RBCs) salvaged during spinal deformity surgery has never been rigorously evaluated. To characterize the usefulness of intraoperatively salvaged RBCs in spinal deformity surgery. The study team hopes to answer the following questions: 1) What is the quality of RBCs salvaged during spine surgery? 2) Does intraoperatively transfused RBC salvage impact clinical outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Any/all patients undergoing spine surgery who utilizes Cell Saver and has blood to be given back.
* This will include pediatric patients 0-17 as well as adults of any age who have been indicated for surgery.
* Only patients with the capacity to consent will be included.

Exclusion Criteria:

* Patients indicated for spinal surgery without the use of Cell Saver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing any spine surgery that utilizes Cell Saver and has blood to be given back.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Lactate Dehydrogenase (LDH) Levels | Day 1 (Day of Surgery)
  LDH assays will be performed following a standardized mechanical stress test will be used to determine whether salvaged red blood cells exhibit signs of fragility ex vivo.
Hemoglobin Levels | Day 1 (Day of Surgery)
  Hemoglobin assays will be performed following a standardized mechanical stress test will be used to determine whether salvaged red blood cells exhibit signs of fragility ex vivo.
Elongation Index (Deformability) | Day 1 (Day of Surgery)
  Ektacytometry will be employed to measure elongation index of salvaged RBCs.
Critical Shear Stress (Aggregation) | Day 1 (Day of Surgery)
  Ektacytometry will be employed to measure critical shear stress of salvaged RBCs.

SECONDARY OUTCOMES:
Standardized Quantified Blood Loss (mL) | Day 1 (Day of Surgery)
Use of Cell Saver | Day 1 (Day of Surgery)
  This will be reported in a binary manner: 0 = yes, 1 = no
Volume (mL) collected via Cell Saver | Day 1 (Day of Surgery)
Units of autologous blood transfused intraoperatively | Day 1 (Day of Surgery)
Units of allogeneic blood transfused intraoperatively | Day 1 (Day of Surgery)
Units of allogeneic blood transfused postoperatively | Day 1 (Day of Surgery)
Duration of pressor use | 1 Day (Day of Surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Lau, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurland DB, Alber D, Smith A, Ahmed S, Orringer D, Frempong-Boadu A, Lau D. What Are We Transfusing? Evaluating the Quality and Clinical Utility of Intraoperatively Salvaged Red Blood Cells in Spinal Deformity Surgery: A Nonrandomized Controlled Trial. Neurosurgery. 2024 Nov 1;95(5):976-985. doi: 10.1227/neu.0000000000003131. Epub 2024 Aug 1. PMID 39087785